CLINICAL TRIAL: NCT02933996
Title: Improvement of Postoperative Immunosuppression in Patients Receiving Coronary Artery Bypass Grafting by Transcutaneous Electrical Acupoint Stimulation: Study Protocol for a Double-blind Randomized Controlled Trial
Brief Title: Improvement of Postoperative Immunosuppression in Patients Receiving Coronary Artery Bypass Grafting by TEAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jiangang Song, deputy director of anesthesia, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14401932600
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Immunosuppression
Keywords: immunosuppression; cardiac surgery; TEAS(Transcutaneous electrical acupoint stimulation); postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAS+GA group (Experimental): The patients of TEAS+GA group will receive TEAS therapy in perioperative period.
  GA: general anesthesia
  Interventions: Device: TEAS+GA group; Device: Sham TEAS+GA group
- Sham TEAS+GA group (Sham Comparator): The patients of Sham TEAS+GA will receive none TEAS in perioperative period.
  Interventions: Device: TEAS+GA group; Device: Sham TEAS+GA group

INTERVENTIONS:
Device: TEAS+GA group — The acupoints including Zusanli and Shenshu, were identified before electrical stimulation with surface electrodes. Selection of these acupoints was based on a consensus between the acupuncturists of the study.
Device: Sham TEAS+GA group — No electrical stimulation sensation is performed in the Sham TEAS group. In the Sham TEAS group, pseudo-stimulation is provided by deliberately connecting the electrodes to the incorrect output socket of the electroacupuncture device, and thus there is no flow of electric current. Patients could see the output light flashing but no current was transmitted throughout the procedure. Patients would be told that the stimulation frequency selected was not perceivable by human beings.

SUMMARY:
The coronary artery bypass grafting (CABG) is a surgery to relieve angina and reduce mortality of coronary heart disease. However, the patient is more prone to have immunosuppression after the surgery, causing secondary infection, and it is closely correlated to the occurrence and progress of tumor after surgery. More and more studies revealed that needle puncture was able to effectively regulate the function of immune system. However, its perioperative application is unclear. Therefore, this clinical study is aimed to evaluate whether the effect of transcutaneous acupoint electric stimulation (TEAS) on improvement of immunosuppression of patients after receiving CABG.

DETAILED DESCRIPTION:
This clinical study was a single-center clinical trial. The 88 patients scheduled to receive CABG under CPB were randomized into 2 groups: the group of TEAS, and the group of transcutaneous acupoint pseudo - electric stimulation (Sham TEAS). Monocytic HLA-DR expression serves as a primary endpoint, and other laboratory parameters (e.g. IL-6, IL-10) and clinical outcomes (e.g. postoperative infectious complications, ICU stay time, and mortality) as the secondary endpoints. In addition, some immune indicators, such as high mobility group protein 1 (HMGB1) and regulatory T cell (Treg), possibly related to the mechanism of TEAS, will also be measured.

This study is a preliminary, mono-center, double-blind, randomized and controlled clinical trial (number of sample, n=88) to explore the effects of TEAS therapy on improvement of postoperative immunosuppression indicated by diminished HLA-DR expression of patients receiving CABG (Fig. 1). The trial will be commenced after ethical approval has been obtained from the Ethics Committee of Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine. All study-related procedures will be performed only after subjects have given their written informed consent. The trial is designed following the Consolidated Standards of Reporting Trials (CONSORT) guidelines, the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) Checklist (Additional file 1), and Standards for Reporting Interventions in Controlled Trials of Acupuncture (STRICTA) recommendations.

We calculate the sample size from the pilot study in our hospital based on the primary outcome Human leukocyte antigen of monocyte (mHLA-DR). In the study, the expression of mHLA-DR three days after surgery was (36.17±5.42) % in the TEAS group and (27.33±3.50) % in the Sham TEAS group, with a power of 80% and 5% Type I error rate. Assuming that the dropout rate to be 10%, 88 patients (n=44 for each group) are needed.

Patients will be recruited from the department of Thoracic and Cardiovascular surgery, at Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine. Potentially eligible subjects who have scheduled for CABG under CPB for coronary diseases will be invited to participate. Patients will be referred from a cardiothoracic surgeon, and then a research assistant will approach the subjects in the general ward pre operation. Patients will be screened and consented for the study. Following the consent, eligible participants will be block randomized into two groups: ⑴ TEAS group (n=44) and ⑵ sham TEAS group (n=44). All patients will conduct a standard operative procedure and postoperative analgesia management. The patients of TEAS group will receive TEAS therapy in perioperative period, and the Sham TEAS will not be performed to receive electrical stimulation sensation in perioperative period. Assessments will be conducted during the perioperative period until 30 days after surgery.

ELIGIBILITY:
Inclusion criteria

1. Aged 18-75 years, male and female;
2. Patients diagnosed as coronary disease, scheduled to receive CABG;
3. BMI: 18.5kg/m2<BMI≤30kg/m2；
4. Graded as I-III by American Standards Association(ASA);
5. Patients firstly receiving CABG under extracorporeal circulation.

Exclusion Criteria

1. Presence of surgical incision or scar at Zusanli acupoint (ST36) /Shenshu (BL23) acupoint;
2. Patients with local skin infection at acupoint;
3. Patients with nerve injury on upper or lower limbs;
4. Patients with history of spinal surgery;
5. Patients who have participated in other clinical trial in recent 4 weeks;
6. Patients using pacemaker;
7. Patients combined with pain before surgery who are using central analgesic drug or drug abuser (e.g., opioid) and dependent user;
8. Patients combined with severe central nervous system disease or severe mental disease;
9. Patients with alcoholic history;
10. Patients who have received emergent coronary bypass operation due to acute myocardial infarction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of mHLA-DR positive cell | day before surgery, Day 1 after surgery (one day after surgery), Day 3 after surgery (3 days after surgery), and Day 5 after surgery (5 days after surgery).
  Human leukocyte antigen of monocyte (mHLA-DR)

SECONDARY OUTCOMES:
Content of serum IL-6 | One day before surgery, Day 1, 3 and 5 after surgery
  interleukin-6 (IL-6)
Content of serum CRP | One day before surgery, Day 1, 3 and 5 after surgery
  reactive protein C (CRP)
Rate of secondary infection | Within 7 days after surgery
  observe the incidence of incision infection, lung infection, hematogenous infection and indwelled catheter infection after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianggang Song, M.D., Principal Investigator — Shuguang Hospital Affiliated to Shanghai University of TCM
Locations (1):
- Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available with 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an extemal independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Chen WT, Wei JF, Wang L, Zhang DW, Tang W, Wang J, Yong Y, Wang J, Zhou YL, Yuan L, Fu GQ, Wang S, Song JG. Effects of perioperative transcutaneous electrical acupoint stimulation on monocytic HLA-DR expression in patients undergoing coronary artery bypass grafting with cardiopulmonary bypass: study protocol for a double-blind randomized controlled trial. Trials. 2019 Dec 30;20(1):789. doi: 10.1186/s13063-019-3889-z. PMID 31888744